CLINICAL TRIAL: NCT00226356
Title: Phase 4 Study: An Open Study of the Efficacy and Tolerability in Unipolar Depression of Augmentation of the One-carbon Cycle With L-methionine, Betaine and Folate
Brief Title: Natural Supplements for Unipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-0048/04/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder | interventions — Betaine; Folic Acid

ARMS (1):
- Supplements of L-methionine, betaine and folate (Experimental)
  Interventions: Drug: Supplements of L-methionine, betaine and folate

INTERVENTIONS:
Drug: Supplements of L-methionine, betaine and folate

SUMMARY:
This study is being conducted to determine the clinical response rate for the regimen of L-methionine, betaine and folate for unipolar depression.

DETAILED DESCRIPTION:
The study is 6 weeks long, with 9 clinical visits. All visits will take place at our location in Massachusetts.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of a MDD or DDNOS; clinical indication for treatment of current depressive symptoms; HDS > 18; women of reproductive potential must use an acceptable method of birth control

Exclusion Criteria:

* Treatment with another psychotropic drug; history of mania or hypomania; history of bipolar illness in first-degree relatives; active homicidality; pregnant; trying to become pregnant, or nursing; unstable medical condition; current substance abuse in the past month; history of sulfa allergy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2007-06 (Actual); Study Completion 2008-09-17 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Dunn, MD, PhD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States